CLINICAL TRIAL: NCT06210347
Title: Patterns of Relapse After Neoadjuvant Chemotherapy in Breast Cancer and Implications for Follow up in Clinical Practice
Brief Title: Patterns of Relapse After Neoadjuvant Chemotherapy in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nour Salah Khairallah, Patterns of Relapse After Neoadjuvant Chemotherapy in Breast Cancer and Implications for Follow up in Clinical Practice, Assiut University
Other Study IDs: breast cancer and NAC
Record Dates: First submitted 2024-01-07; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to identify patterns of relapse after Neoadjuvant Chemotherapy (NAC) for breast cancer to refine follow up recommendations.

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy (NAC) is usually used to facilitate breast-conserving surgery and improve surgical outcomes for breast cancer patients [1]. In addition, NAC can help to eradicate micrometastatic disease and serve to test chemosensitivity while providing similar survival benefits to adjuvant chemotherapy [2-5] .

Pathologic complete response (pCR) after neoadjuvant chemotherapy is associated with superior survival outcomes, with higher rates of pCR in human epidermal growth factor receptor 2 positive (HER2+) and triple negative breast cancer (TNBC) subtypes compared to hormone receptor (HR)-positive subtypes [6-7] .

Patients who achieve pCR also remain at signifcant risk of relapse, with studies reporting 5-year disease-free survival (DFS) rates of 75-87% [2,8-10] . Retrospective study of 88 Japanese patients who achieved pCR reported a recurrence rate of 13.6% and all relapses occurred within 32 months from diagnosis [11].

There for, little is known about the patterns of relapse after NAC especially in the real world. There are currently no specific guidelines for post-treatment follow-up of patients treated with NAC and variations in practice exist. So, this study aims to evaluate the relapse risks in different subgroups of breast cancers treated with NAC and determine the associated time trends and patterns of relapse in these patients. These findings may potentially lead to the development of risk-adapted surveillance strategies for patients treated with NAC

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged >= 18
2. Pathologically proved breast cancer
3. PS 0-1 (ECOG)
4. Patients indicated to receive NAC

Exclusion Criteria:

1. Patients with metastatic disease at diagnosis
2. Patients who did not undergo subsequent curative intent surgery
3. Those who received Neoadjuvant hormonal treatment
4. Those that had incomplete treatment information

Ages: 18 Years to 100 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study will be carried out at SECI between 2018 and 2022 . All cases with inclusion criteria will be included .
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
The patterns of relapse after Neoadjuvant Chemotherapy (NAC) for breast cancer to refine follow up recommendations. | 2 years
  Patterns of relapse after Neoadjuvant Chemotherapy (NAC) in breast cancer patients to refine follow up recommendations.

REFERENCES:
- [Background] Fisher B, Bryant J, Wolmark N, Mamounas E, Brown A, Fisher ER, Wickerham DL, Begovic M, DeCillis A, Robidoux A, Margolese RG, Cruz AB Jr, Hoehn JL, Lees AW, Dimitrov NV, Bear HD. Effect of preoperative chemotherapy on the outcome of women with operable breast cancer. J Clin Oncol. 2023 Apr 1;41(10):1795-1808. doi: 10.1200/JCO.22.02571. PMID 36989610
- [Background] van der Hage JA, van de Velde CJ, Julien JP, Tubiana-Hulin M, Vandervelden C, Duchateau L. Preoperative chemotherapy in primary operable breast cancer: results from the European Organization for Research and Treatment of Cancer trial 10902. J Clin Oncol. 2001 Nov 15;19(22):4224-37. doi: 10.1200/JCO.2001.19.22.4224. PMID 11709566
- [Background] Mauri D, Pavlidis N, Ioannidis JP. Neoadjuvant versus adjuvant systemic treatment in breast cancer: a meta-analysis. J Natl Cancer Inst. 2005 Feb 2;97(3):188-94. doi: 10.1093/jnci/dji021. PMID 15687361
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Long-term outcomes for neoadjuvant versus adjuvant chemotherapy in early breast cancer: meta-analysis of individual patient data from ten randomised trials. Lancet Oncol. 2018 Jan;19(1):27-39. doi: 10.1016/S1470-2045(17)30777-5. Epub 2017 Dec 11. PMID 29242041
- [Background] Kong X, Moran MS, Zhang N, Haffty B, Yang Q. Meta-analysis confirms achieving pathological complete response after neoadjuvant chemotherapy predicts favourable prognosis for breast cancer patients. Eur J Cancer. 2011 Sep;47(14):2084-90. doi: 10.1016/j.ejca.2011.06.014. Epub 2011 Jul 5. PMID 21737257
- [Background] Cortazar P, Zhang L, Untch M, Mehta K, Costantino JP, Wolmark N, Bonnefoi H, Cameron D, Gianni L, Valagussa P, Swain SM, Prowell T, Loibl S, Wickerham DL, Bogaerts J, Baselga J, Perou C, Blumenthal G, Blohmer J, Mamounas EP, Bergh J, Semiglazov V, Justice R, Eidtmann H, Paik S, Piccart M, Sridhara R, Fasching PA, Slaets L, Tang S, Gerber B, Geyer CE Jr, Pazdur R, Ditsch N, Rastogi P, Eiermann W, von Minckwitz G. Pathological complete response and long-term clinical benefit in breast cancer: the CTNeoBC pooled analysis. Lancet. 2014 Jul 12;384(9938):164-72. doi: 10.1016/S0140-6736(13)62422-8. Epub 2014 Feb 14. PMID 24529560
- [Background] Tanioka M, Shimizu C, Yonemori K, Yoshimura K, Tamura K, Kouno T, Ando M, Katsumata N, Tsuda H, Kinoshita T, Fujiwara Y. Predictors of recurrence in breast cancer patients with a pathologic complete response after neoadjuvant chemotherapy. Br J Cancer. 2010 Jul 27;103(3):297-302. doi: 10.1038/sj.bjc.6605769. Epub 2010 Jul 6. PMID 20606681
- [Background] Wolmark N, Wang J, Mamounas E, Bryant J, Fisher B. Preoperative chemotherapy in patients with operable breast cancer: nine-year results from National Surgical Adjuvant Breast and Bowel Project B-18. J Natl Cancer Inst Monogr. 2001;(30):96-102. doi: 10.1093/oxfordjournals.jncimonographs.a003469. PMID 11773300